CLINICAL TRIAL: NCT02570399
Title: Feasibility Study of High Dose Stereotactic Body Radiation Therapy (SBRT) for Lymph Nodal Lesions in Oligometastatic Patients for Genito-urinary, Gastro-intestinal and Gynaecological Cancer
Brief Title: High Dose SBRT for Abdominal-Pelvic Lymph Nodal Lesions in Oligometastatic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Principal Investigator, Michele Tedeschi, MD, Istituto Clinico Humanitas
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1388
Record Dates: First submitted 2015-09-28; First posted 2015-10-07 (Estimated); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Lymph Node Cancer Metastatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lymph nodal metastatic lesions (Experimental): Oligometastatic patients with abdominal-pelvic lymph nodes
  Interventions: Radiation: Oligometastatic patients with abdominal-pelvic lymph nodes

INTERVENTIONS:
Radiation: Oligometastatic patients with abdominal-pelvic lymph nodes — Hypofractionated ablative radiation therapy for oligometastatic patients with lymph node metastases

SUMMARY:
This is a prospective, multicentric, phase II and feasibility study aimed to address early and late side effects of hypofractionated ablative radiotherapy for oligometastatic patients with lymph node metastases for genito-urinary, gastro-intestinal and gynaecological cancer.

DETAILED DESCRIPTION:
The purpose of this prospective, multicentric, phase II study is to determine the feasibility of Stereotactic Body Radiation Therapy in stage IV selected oligometastatic patients, by looking at acute and late toxicity. Investigators also want to verify what is the impact of local control in irradiated metastatic foci in the context of the systemic disease, how local control can affect disease free survival and overall survival, and moreover quality of life of patients treated.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* WHO performance status ≤ 2
* Histologically-proven of primary cancer disease
* M1 stage with primary cancer site radically treated with complete response/resection or stable. No other site of disease in progression (a maximum of 3 lymph node sites of disease to treat)
* Diameter ≤ 5 cm
* Abdomen/pelvic site
* Informed consent.

Exclusion Criteria:

* Patients were required to have not brain metastases or bone metastases.
* Patients with a life expectancy of >3 months.
* Any serious disease contraindicated radiation therapy
* Other coexisting malignancies, uncontrolled intercurrent illness, active infectious processes, and exudative, bloody, or cytologically malignant effusions excluded patients from the trial. Additionally, patients were excluded from the trial if they were receiving any systemic chemotherapy during radiotherapy, although hormonal therapy was allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2015-02-26 (Actual); Primary Completion 2019-03-26 (Actual); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility in terms of toxicity related to radiation therapy | 2 months
  Evaluation of acute and late toxicity performed during and after radiation therapy

SECONDARY OUTCOMES:
Tumour response to local radiation therapy (RECIST criteria) | 2 months
  Evaluation of tumour response to local radiation therapy by means of imaging
Overall survival in the oligometastatic patients | 2 months
  Statistical evaluation of how local control of the metastatic disease can affect overall survival
Disease free survival in the oligometastatic patients | 2 months
  Statistical evaluation of how local control of the metastatic disease can affect disease free survival
Quality of life questionnaire of treated patients | 2 months
  Evaluation of quality of life of patients during and after radiation therapy

CONTACTS AND LOCATIONS:
Overall Officials: Ciro Franzese, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milano, Italy

REFERENCES:
- [Derived] Franzese C, Comito T, Tripoli A, Franceschini D, Clerici E, Navarria P, Badalamenti M, D'agostino G, Loi M, Mancosu P, Reggiori G, Tomatis S, Scorsetti M. Phase II trial of high dose stereotactic body radiation therapy for lymph node oligometastases. Clin Exp Metastasis. 2020 Oct;37(5):565-573. doi: 10.1007/s10585-020-10047-x. Epub 2020 Jun 15. PMID 32556682